CLINICAL TRIAL: NCT07384013
Title: Impact of Metamizole (Optalgin®) on Anti-Xa Concentrations in Oncology Patients Receiving DOACs
Brief Title: Study Protocol: Impact of Metamizole (Optalgin®) on Anti-Xa Concentrations in Oncology Patients Receiving DOACs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0268-25-RMB
Record Dates: First submitted 2025-09-25; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Oncologic Diseases; Coagulation Defect; Pain Management
Keywords: Direct Oral Anticoagulants (DOACs); Optalgin
MeSH Terms: conditions — Hemostatic Disorders; Agnosia | interventions — Dipyrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Chronic metamizole users (Experimental): Patients receiving Optalgin prior to study enrollment
  Interventions: Drug: metamizole
- Cohort 2: New metamizole users (Experimental): Patients receiving Optalgin after to study enrollment
  Interventions: Drug: metamizole

INTERVENTIONS:
Drug: metamizole — chronic metamizole use
  Other Names: OPTALGIN
Drug: metamizole — New metamizole users

SUMMARY:
Evaluation of the Effect of metamizole (Optalgin®) on Anti-Xa Levels in Oncology Patients Receiving Direct Oral Anticoagulants (DOACs)

DETAILED DESCRIPTION:
Evaluation of the Effect of metamizole (Optalgin®) on Anti-Xa Levels in Oncology Patients Receiving Direct Oral Anticoagulants (DOACs)

ELIGIBILITY:
Inclusion Criteria:

* Adult oncology patients (≥18 years old).
* Receiving apixaban or rivaroxaban for anticoagulation.
* New/current metamizole users taking at least 1g TID for pain management.
* Platelets ≥100×10⁹/L
* ECOG PS<3
* Provided informed consent

Exclusion Criteria:

* History of allergic reaction to metamizole or DOACs.
* Individuals with significant gastrointestinal disorders that may affect absorption, including (but not limited to) diagnosed bowel obstruction, persistent diarrhea, or the presence of a nasogastric tube (NGT/zonda)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in DOAC | 1- Baseline 2- End Of Treatment 3- Day 3 Post treatment 4- Day 5 Post Treatment 5- Day 7 Post treatment
  Change in DOAC peak and trough concentrations during periods with and without metamizole comedication (5 different time points).

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided